CLINICAL TRIAL: NCT05324930
Title: Evaluating the Effectiveness of Collagen Matrix Dressing on Neuropathic Diabetic Foot Ulcer in T2DM Patients: a Randomised Control Trial
Brief Title: Evaluating the Effectiveness of Piscean Derived Collagen Dressing on Neuropathic Diabetic Foot Ulcer in T2DM Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Dr Zainab Khan, Chief Resident, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDDF37628
Record Dates: First submitted 2022-04-01; First posted 2022-04-13 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Foot Ulcer Neuropathic; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized control trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients were randomized, all boxes of dressings were opened and healthcare professional applying the dressing and assessing the wound was unaware of what treatment is being given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): After conventional therapy consisting of debridement, infection control and offloading, patients received a saline-moistened gauze dressing (control group) for wound care.
  Interventions: Device: Saline infused dressing
- Experimental group (Experimental): After conventional therapy consisting of debridement, infection control and offloading, patients received the piscean collagen dressing (the study group) for wound care.
  Interventions: Device: Piscean collagen dressing

INTERVENTIONS:
Device: Piscean collagen dressing — Piscean collagen dressing
  Other Names: Dressing
  Arms: Experimental group
Device: Saline infused dressing — Saline infused dressing
  Arms: Control group

SUMMARY:
Diabetic foot ulcers (DFU) are challenging to treat with complicated healing processes and require advanced wound care. Piscean collagen has the potential to promote the regenerative process while remaining cost-effective and with minimal side effects. In this study, the efficacy of a piscean collagen matrix dressing was compared with a standard dressing of saline-moistened gauze for wound healing in patients with neuropathic DFU.

This is a double-blinded, randomised clinical trial.

DETAILED DESCRIPTION:
Diabetic foot ulcers (DFU) are challenging to treat with complicated healing processes and require advanced wound care. Piscean collagen has the potential to promote the regenerative process while remaining cost-effective and with minimal side effects. In this study, the efficacy of a piscean collagen matrix dressing was compared with a standard dressing of saline-moistened gauze for wound healing in patients with neuropathic DFU.

This is a double-blinded, randomised clinical trial. After conventional therapy consisting of debridement, infection control and offloading, patients were randomly allocated to receive either a piscean matrix dressing (the study group) or a saline-moistened gauze dressing (control group) for wound care. The reduction in DFU size and the number of patients with complete healing were measured throughout the treatment and in follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients with neuropathic DFUs at Grades I or II for a period of at least 12 weeks, based on the Wagner classification;
* be able to understand simple instructions and provided voluntary, signed informed consent.

Exclusion Criteria:

* active infection which might lead to hospitalisation, gangrene,
* systemic inflammatory or autoimmune disease
* renal failure
* presence of ischaemia or osteomyelitis

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in DFU size | 3 months
  change in DFU size using the manual planimetric method

SECONDARY OUTCOMES:
Complete wound healing | 3 months
  Complete wound healing using three-dimensional wound measurement software

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Khan, MD, Principal Investigator — Punjab Care hospital
Locations (1):
- Zainab Khan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be provided upon reasonable request